CLINICAL TRIAL: NCT02629497
Title: Role of 12-lipoxygenase in Platelet Reactivity and Type 2 Diabetes Mellitus
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Michael Holinstat, Associate Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HL 114405; R01HL114405 (NIH); ODS (Other: Office of Dietary Supplementation (NIH), co-funder)
Record Dates: First submitted 2015-01-14; First posted 2015-12-14 (Estimated); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Thrombosis; Type 2 Diabetes Mellitus
Keywords: platelets; 12-lipoxygenase; fatty acids; DGLA; DHA; EPA; 12-LOX
MeSH Terms: conditions — Thrombosis; Diabetes Mellitus, Type 2 | interventions — evening primrose oil; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Healthy subjects for Omega-6 protection (Experimental): Platelets from healthy donors will be assessed for regulation by Primrose Oil (omega-6 fatty acid).
  Interventions: Dietary Supplement: Primrose oil
- T2DM patients for Omega-6 protection (Experimental): platelets from Type 2 diabetes mellitus (T2DM) patients will be assessed for regulation by Primrose Oil (omega-6 fatty acid).
  Interventions: Dietary Supplement: Primrose oil
- Healthy control for Omega-3 protection (Active Comparator): Platelets from healthy donors will be assessed for regulation by Fish Oil (omega-3 fatty acid).
  Interventions: Dietary Supplement: Fish Oil
- T2DM for Omega-3 protection (Active Comparator): platelets from Type 2 diabetes mellitus (T2DM) patients will be assessed for regulation by Fish Oil (omega-3 fatty acid).
  Interventions: Dietary Supplement: Fish Oil

INTERVENTIONS:
Dietary Supplement: Primrose oil — T2DM patients and matched controls subjects will be given Primrose oil for 2 months, followed by 2-week washout. Blood will be drawn at the beginning, during, and following treatments and platelet function will be assessed.
  Arms: Healthy subjects for Omega-6 protection; T2DM patients for Omega-6 protection
Dietary Supplement: Fish Oil — T2DM patients and matched controls subjects will be given Fish oil for 2 months, followed by 2-week washout. Blood will be drawn at the beginning, during, and following treatments and platelet function will be assessed.
  Other Names: DHA/EPA
  Arms: Healthy control for Omega-3 protection; T2DM for Omega-3 protection

SUMMARY:
This study investigates the potential protective effects of fatty acid supplementation through inhibition of platelet activation. fatty acids (omega-3 and omega-6) will be evaluated for protection from agonist-mediated platelet activation in platelets from type 2 diabetics and healthy controls. Post-menopausal women with type 2 diabetes mellitus and healthy post-menopausal women will be treated with omega-3 and omega-6 fatty acid supplements to determine protection from platelet activation and thrombosis in this high risk population.

DETAILED DESCRIPTION:
Essential fatty acids such as omega-3 and omega-6 have been shown to play important roles in regulating platelet activation, but the underlying mechanisms have not been fully elucidated as well as their true protection from thrombosis.

12-lipoxygenase oxidized fatty acids are known to play both a pro- and anti-thrombotic effect on platelets depending on the fatty acid. oxidation of arachidonic acid by 12-lipoxygenase resuts in a pro-thrombotic bioactive lipid whereas oxidation of the omega-6 fatty acid DGLA found in plant oil results in formation of a potent anti-thrombotic bioactive lipid. Determining the extent of protection from this and other bioactive lipids produced through oxygenase activity will allow for a better understanding of which fatty acid supplementation may best protect from thrombosis.

Essential fatty acids such as omega-3 (DHA/EPA) and omega-6 (DGLA) appear to be protective. However the underlying mechanism for this potential protection is not well understood. Identifying the mechanism by which these supplements protect from platelet activation may identify new approaches to preventing thrombotic events in this high risk population.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects and T2DM patients
* Postmenopausal women with T2DM
* All races and ethnicities
* T2DM patients taking 1st line diabetic treatment (i.e. Metformin)

Exclusion Criteria:

* Fish and plant oil supplements 2 months prior to enrollment
* NSAIDS and aspirin 1 week prior to enrollment
* Cardiovascular event within 6 months prior to enrollment
* Other anti-platelet treatment including PDE and P2Y12 inhibitors

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-11; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
platelet reactivity | through study completion, an average of 1 year
  decreased platelet activity ex vivo translating to protection from clot formation in vivo

SECONDARY OUTCOMES:
fatty acid incorporation | through study completion, an average of 1 year
  measure altered levels of essential fatty acids in blood and platelets following treatment
Oxylipin production | through study completion, an average of 1 year
  determine the oxylipin products formed following each intervention

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Holinstat, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yamaguchi A, Stanger L, Freedman JC, Prieur A, Thav R, Tena J, Holman TR, Holinstat M. Supplementation with omega-3 or omega-6 fatty acids attenuates platelet reactivity in postmenopausal women. Clin Transl Sci. 2022 Oct;15(10):2378-2391. doi: 10.1111/cts.13366. Epub 2022 Jul 25. PMID 35791734